CLINICAL TRIAL: NCT07344675
Title: Relationship Between Fibromyalgia Syndrome and Chronic Pelvic Pain: A Cross-Sectional Study
Brief Title: Fibromyalgia Syndrome and Chronic Pelvic Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 4926 (June 17, 2025)
Record Dates: First submitted 2026-01-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Fibromyalgia Syndrome; Pain; Chronic Pelvic Pain; Chronic Pelvic Pain Syndrome (CPPS)
Keywords: fibromyalgia; chronic pelvic pain; pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Those with fibromyalgia syndrome: Female patients with a history of follow-up and treatment due to fibromyalgia syndrome
- Female patients presenting to the outpatient clinic who do not have fibromyalgia syndrome: Patients who do not have a history of fibromyalgia syndrome and who present to the outpatient clinic for other reasons

SUMMARY:
This study aimed to compare patients with and without fibromyalgia syndrome in terms of chronic pelvic pain and pelvic floor dysfunction.

DETAILED DESCRIPTION:
The study planned for two patient groups in the Physical Medicine and Rehabilitation outpatient clinic: female patients followed up for fibromyalgia and a control group matched for age and gender without fibromyalgia syndrome. Demographic data, symptom duration, chronic pelvic pain, and pelvic dysfunction symptoms will be assessed in both groups. Pain levels will be measured using the Visual Analog Scale and the McGill Pain Questionnaire Short Form. Additionally, the Fibromyalgia Impact Questionnaire, the Chronic Pelvic Pain Impact Questionnaire, and the Short Form-12 for quality of life assessment will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 and over
* Voluntary participation in the study

Exclusion Criteria:

* Individuals with cognitive impairment
* History of pelvic surgery within the last 3 months
* Severe cardiac, renal, liver disease, respiratory or endocrine dysfunction, uncontrolled psychiatric illness
* Pregnant or breastfeeding women
* Individuals with neuropathy or central nervous system disorders
* History of neoplasm in the pelvic region

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female participants aged 18 and over, with and without fibromyalgia syndrome
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Day 1
  The score is obtained by measuring, with a ruler, the distance in millimeters along the 10-cm line from the "no pain" reference point to the mark indicated by the patient, yielding a total score between 0 and 100, where higher values reflect increased pain severity.
Short-Form McGill Pain Questionnaire | Day 1
  The Short-Form McGill Pain Questionnaire was developed as a condensed version of the original instrument. Its core section includes 15 pain descriptors, consisting of 11 sensory and 4 affective items, each rated according to intensity on a 4-point scale from 0 (no pain) to 3 (severe pain).
Pelvic Pain Impact Questionnaire | Day 1
  The self-administered Pelvic Pain Impact Questionnaire assesses the effect of pelvic pain on daily life. It comprises 8 mandatory and 2 optional items, each rated on a 5-point Likert scale, yielding a total score from 0 to 32, with higher scores indicating greater impact on daily functioning.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Day 1
  The Fibromyalgia Impact Questionnaire (FIQ) is a self-administered tool consisting of 10 items; the first item includes 11 questions assessing physical functioning, each rated on a 4-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided